CLINICAL TRIAL: NCT07380087
Title: Efficacy of Suprascapular Nerve Block on the Tolerability and Effectiveness of Shoulder Hydrodistension in Patients With Adhesive Capsulitis: A Randomized Clinical Trial
Brief Title: Suprascapular Nerve Block to Improve Tolerance and Outcomes of Shoulder Hydrodistension in Adhesive Capsulitis
Acronym: SHINE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, João Rocha Neves, MD, MSc, MPH, PhD, MBA, FEBVS, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMUP/ULSSJ - 01/2026
Record Dates: First submitted 2026-01-18; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Adhesive Capsulitis; Adhesive Capsulitis of Unspecified Shoulder; Adhesive Capsulitis, Shoulder; Frozen Shoulder; Shoulder Pain; Shoulder Stiffness
Keywords: Shoulder Hydrodistension; Suprascapular Nerve Block; Shoulder Pain; Shoulder Mobility; Randomized Clinical Trial; Pain Management; Rehabilitation
MeSH Terms: conditions — Bursitis; Shoulder Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-group randomized clinical trial comparing hydrodistension alone versus suprascapular nerve block followed by hydrodistension in patients with adhesive capsulitis. Participants are allocated in a 1:1 ratio using a pre-generated randomization sequence. Both groups undergo a single intervention session, with outcomes assessed at baseline, 1 month, and 3 months.
Masking Description: This is an open-label study. No participants, care providers, or outcome assessors are masked, and no additional masking procedures are used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrodistension Alone (Active Comparator): Participants assigned to this arm will undergo standard ultrasound-guided shoulder hydrodistension without any prior nerve block. The procedure consists of an anterior intra-articular injection of 20 mL of normal saline, 4 mL of ropivacaine, and 40 mg of methylprednisolone. This intervention represents the current standard treatment for adhesive capsulitis.
  Interventions: Procedure: Shoulder Hydrodistention
- Suprascapular Nerve Block Followed by Shoulder Hydrodistension (Experimental): Participants in this arm will receive an ultrasound-guided suprascapular nerve block immediately before the hydrodistension procedure. The nerve block is performed at the suprascapular notch using 2 mL of ropivacaine. After the block, participants undergo standard anterior shoulder hydrodistension consisting of an intra-articular injection of 20 mL of normal saline, 4 mL of ropivacaine, and 40 mg of methylprednisolone. This combined approach is intended to improve procedural tolerance and potentially enhance clinical outcomes in adhesive capsulitis.
  Interventions: Procedure: Shoulder Hydrodistention; Procedure: suprascapular nerve block

INTERVENTIONS:
Procedure: Shoulder Hydrodistention — Shoulder hydrodistension is performed using an anterior intra-articular approach. The procedure consists of an injection of 20 mL of normal saline, 4 mL of ropivacaine, and 40 mg of methylprednisolone into the glenohumeral joint, with the aim of capsular distension, pain reduction, and improvement of shoulder mobility.
  Other Names: Hydrodilation; Glenohumeral Hydrodistension
Procedure: suprascapular nerve block — The suprascapular nerve block is performed under ultrasound guidance at the suprascapular notch using an injection of 2 mL of ropivacaine. The block is administered immediately before shoulder hydrodistension with the aim of reducing procedural pain and improving patient tolerance.
  Other Names: Suprascapular Block; SSNB
  Arms: Suprascapular Nerve Block Followed by Shoulder Hydrodistension

SUMMARY:
Adhesive capsulitis ("frozen shoulder") causes significant pain and loss of shoulder mobility. Shoulder hydrodistension is an established treatment that can improve movement and reduce symptoms, but the procedure itself may be painful and difficult for some patients to tolerate.

This randomized clinical trial will evaluate whether performing a suprascapular nerve block with local anesthetic immediately before hydrodistension can reduce pain during the procedure, improve patient comfort, and potentially enhance clinical outcomes.

Participants will be randomly assigned to one of two groups:

hydrodistension alone, or

suprascapular nerve block followed by hydrodistension.

Pain, shoulder mobility, functional ability, psychological measures, and quality of life will be assessed at baseline, 1 month, and 3 months after the procedure. The study aims to determine whether adding a suprascapular nerve block provides better tolerability and improved recovery for patients with adhesive capsulitis.

DETAILED DESCRIPTION:
1 Efficacy of suprascapular nerve block on the tolerability and efficacy of shoulder hydrodistension in patients with adhesive capsulitis: randomized clinical trial

* Principal Investigator Name: João Paulo Castro Contact: jpcastro@med.up.pt

  Under the supervision of:

  Professor José Paulo Andrade Full Professor at the Faculty of Medicine of the University of Porto Professor Iva Brito Senior Consultant in Rheumatology at the Local Health Unit of São João EPE and Invited Professor at the Faculty of Medicine of the University of Porto

  Porto - January 2026

  Identification of the Research Unit Physical Medicine and Rehabilitation Service of the Local Health Unit of São João, EPE

  ________________________________________
* Scientific justification and context Adhesive capsulitis of the shoulder is a frequent pathology, characterized by pain and progressive limitation of joint mobility, with a significant impact on the quality of life and functionality of patients (1). Shoulder joint hydrodistension is considered one of the treatments of choice, demonstrating effectiveness in reducing pain and improving range of motion. However, the procedure can be painful, which may limit its tolerability and potentially the therapeutic aggressiveness required for effective capsular distension (2, 3).

  Suprascapular nerve block, using local anesthetics such as ropivacaine, is a known technique for controlling shoulder pain (4, 5). Its use prior to hydrodistension may:
  * Reduce pain during the procedure
  * Improve patient tolerance
  * Allow greater capsular distension
  * Potentially improve clinical outcomes and prognosis To date, there is limited and heterogeneous evidence on the impact of this block as an adjunct to hydrodistension, justifying the performance of this clinical trial.
* Study Objectives Main Objective To evaluate the evolution of shoulder pain and mobility in patients with adhesive capsulitis undergoing hydrodistension, with or without suprascapular nerve block.

  Pain will be assessed using the Numerical Pain Scale (NRS), and shoulder mobility will be assessed by goniometry of joint ranges of motion.

  Assessments will be conducted at three points in time:
  * Before the procedure (baseline)
  * 1 month after the procedure
  * 3 months after the procedure Secondary objectives

  To evaluate the impact of the intervention on psychological, functional, and quality of life dimensions, namely:
  * Anxiety and depression, assessed using the Hospital Anxiety and Depression Scale (HADS)
  * Kinesiophobia, assessed using the Tampa Scale for Kinesiophobia
  * Health-related quality of life, assessed using the EQ-5D-5L
  * Upper limb functionality, assessed using the QuickDASH and the Shoulder Pain and Disability Index (SPADI)

  These variables will be assessed at two points in time:
  * Baseline
  * 3 months after the procedure Additionally, the need for physiotherapy and its duration after the procedure will be evaluated.
* Study Design

  * Prospective clinical trial
  * Randomized
  * Two parallel arms
  * Open-label
  * Single intervention
* Study Population Inclusion Criteria

  * Adults ≥ 18 years
  * Clinical diagnosis of adhesive capsulitis of the shoulder
  * Persistent pain and functional limitation despite initial conservative treatment
  * Ability to understand and sign informed consent Exclusion Criteria
  * Known allergy to ropivacaine or methylprednisolone
  * Active local or systemic infection
  * Uncontrolled coagulopathy or anticoagulation
  * Recent prior surgery of the affected shoulder
  * Neurological disease affecting the upper limb
  * Pregnancy

  Sample size (calculation and assumptions) Proposed primary endpoint: pain and mobility 3 months after hydrodistension (Numerical Pain Scale, NRS 0-10).

  Clinical hypothesis: suprascapular nerve block reduces pain during the procedure.

  Assumptions for calculation (conservative and clinically plausible):
  * Clinically relevant minimum difference (Δ): 2 points on the VAS
  * Standard deviation (SD): 2.5 (typical variability in procedural pain)
  * Two-tailed test, α = 0.05; Power (1-β) = 80%

  Result of the calculation (comparison of means, 2 groups):
  * Approximately 25 participants per group are needed (total 50) Adjustment for losses/dropouts (≈15%)
  * 25 / (1-0.15) ≈ 29.4 → rounding: 30 per group
  * Proposed final sample size: 60 participants (30+30)
* Randomization

  Participants will be randomly assigned in a 1:1 ratio to:
  * Control Group: Isolated hydrodistension
  * Intervention Group: Suprascapular nerve block followed by hydrodistension Randomization will be performed using a previously generated random sequence.
* Interventions 8.1 Shoulder Hydrodistension (both groups)

  Performed anteriorly, with intracapsular injection of:
  * 20 ml of saline solution
  * 4 ml of ropivacaine
  * 40 mg of methylprednisolone

  8.2 Suprascapular Nerve Block (intervention group)

  Performed prior to hydrodistension, consisting of an injection of:

  • 5 ml of ropivacaine The block will be performed in the suprascapular notch, on the posterior aspect of the shoulder, according to a standardized technique.

  There will be no sham intervention.

  ________________________________________
* Concomitant Treatments Physiotherapy after the procedure is permitted and not restricted by the protocol. In general, the duration of physiotherapy is expected to be shorter after effective hydrodistension.

  ________________________________________
* Outcome Evaluation Evaluation Times

  Outcomes will be evaluated at three distinct times:
  * Before the procedure (baseline)
  * 1 month after the procedure
  * 3 months after the procedure Pain during the procedure will be evaluated exclusively at the time of the clinical act.

  Primary Outcome

  • Pain and mobility, assessed using the Numerical Pain Scale (NRS, 0-10), 3 months after hydrodistension.

  Pain
  * Shoulder pain at rest and/or with movement, as assessed by the Numerical Pain Scale (NRS)
  * Assessed at baseline, 1 month, and 3 months

  Shoulder Mobility
  * Assessment of joint range of motion (flexion, abduction, external rotation, and internal rotation), measured by goniometry
  * Assessed at baseline, 1 month, and 3 months

  Secondary Outcomes Shoulder and Upper Limb Functionality
  * Shoulder Pain and Disability Index (SPADI)
  * Quick Arm, Shoulder, and Hand Disabilities (QuickDASH)
  * Assessed at baseline and at 3 months

  Health-Related Quality of Life
  * Assessed using the EQ-5D-5L
  * Assessed at baseline and at 3 months

  Psychological Dimension
  * Anxiety and depression, assessed using the Hospital Anxiety and Depression Scale (HADS)
  * Kinesiophobia, assessed using the Tampa Scale for Kinesiophobia
  * Assessed at baseline and at 3 months

  Physical Therapy
  * Need for physical therapy after the procedure (yes/no)
  * Duration of physical therapy, measured in number of sessions or weeks of treatment

  Safety

  • Systematic recording of adverse events, including:
  * Prolonged pain
  * Hematoma
  * Infection
  * Transient or persistent neurological deficit
  * Adverse reactions to the drugs used Adverse events will be classified according to severity, causal relationship with the procedure, and need for additional intervention.
* Safety and Risks Risks of hydrodistension

  * Transient pain
  * Hematoma
  * Infection (rare)
  * Adverse drug reactions Additional risks of suprascapular block
  * Local pain or discomfort
  * Hematoma
  * Transient numbness or weakness of the shoulder
  * Accidental vascular puncture
  * Adverse reactions to ropivacaine
  * Nerve injury (extremely rare) All procedures will be performed by an experienced professional, respecting safety and asepsis standards.
* Expected Benefits

  * Possible reduction of pain associated with the procedure
  * Improved tolerability of hydrodistension
  * Potential improvement in clinical outcomes
  * Contribution to scientific knowledge Direct individual benefit is not guaranteed.
* Ethical Considerations

  * Participation is voluntary
  * Participants may leave the study at any time without clinical detriment
  * The study complies with the principles of the Declaration of Helsinki
  * Written informed consent will be obtained before any procedure
* Data Protection and GDPR Data will be processed in accordance with the GDPR Participants will be identified by code Only the research team will have access to identifiable data Data will be used exclusively for scientific purposes Participants may exercise their legal rights over the data at any time The anonymity and confidentiality of participants will be safeguarded. The patient will be entered without any reference to their name. The participant number will correspond to the clinical information in a separate database, which will only be used for the proposed purpose, after supervision by Master João Paulo Castro and the service director. For analysis purposes, the participant number will be deleted.

  All information entered into the database will be recorded in the medical record.

  Rules of Ethical Conduct and Good Practices will be observed to ensure compliance with the precepts of the Declaration of Helsinki, the Convention on Human Rights and Biomedicine, the guidelines of the Council for International Organizations of Medical Sciences, and the Guide to Good Clinical Practices.
* Data Management and Preservation Data will be stored in a secure physical and/or digital medium for the legally required period and subsequently destroyed.

  Patient characterization will be performed, including demographic data, clinical symptoms and associated comorbidities, as well as a description of the surgical techniques used and adverse events that occurred (Appendix 1).

  Data collection will be carried out by Master João Paulo Castro, through clinical interviews and consultation of patient records.

  Statistical data processing will be performed by Master João Paulo Castro. According to the General Data Protection Regulation (GDPR), data collection will be carried out through registration in a protected Excel spreadsheet, and no patient identification data will be transferred. Each participant will be uniquely identified by a code number, which will be subsequently deleted.

  The data will be exported in .xls and .sav formats, compatible with appropriate statistical software, i.e., R, SPSS, Stata, and Microsoft Excel.
* Funding and Conflicts of Interest The study does not involve external funding or known conflicts of interest. No additional costs are foreseen for the Local Health Unit of São João, EPE, beyond the usual study and provision of materials recommended for the treatment of the aforementioned pathologies.

  There will be no abuse of hospital resources or any others, which will be determined by the management of the Physical Medicine and Rehabilitation service.
* Dissemination of results The results may be presented at scientific conferences and published in indexed scientific journals with an impact factor, always guaranteeing the anonymity of the participants.

  ________________________________________
* Schedule (operational estimate) Total estimated duration: ~12 months

1. Preparation and ethical approval (Months 0-2)

* Submission to the Ethics Committee and response to any requests for clarification
* Final versions: Information/Consent Sheet, CRF (case report form) and database 2. Recruitment and inclusion (Months 3-8)
* Consecutive screening of eligible patients in consultation/referral
* Randomization and performance of the procedure (block +/- hydrodistension) 3. Clinical follow-up (Months 3-10)
* Standardized post-procedure assessments at defined times (D0, 1 month and 3 months) 4. Statistical analysis and writing (Months 10-12)
* Closing the database, final analysis, submission to congress/journal

Bibliografia:

1. Brindisino F, Garzonio F, Turolla A, Andriesse A, Pulina F, Cucchi D, et al. Perspectives, perceptions, and expectations of subjects with frozen shoulder: a web-based Italian survey. Arch Physiother. 2024;14:116-30.
2. Konarski A, Narayanasamy K, Coghlan J, Chung T, Andrews M, Bell S. A Double Blind Randomised Controlled Trial Comparing Glenohumeral Cortisone With and Without Hydrodilatation in Patients With Frozen Shoulder. ANZ J Surg. 2025;95(10):2162-70.
3. Wang JC, Tsai PY, Hsu PC, Huang JR, Wang KA, Chou CL, et al. Ultrasound-Guided Hydrodilatation With Triamcinolone Acetonide for Adhesive Capsulitis: A Randomized Controlled Trial Comparing the Posterior Glenohumeral Recess and the Rotator Cuff Interval Approaches. Front Pharmacol. 2021;12:686139.
4. Goffin P, Forthomme B, Lecoq JP, Benmouna K, Kaux JF, Fontaine R. Evaluation of intensive rehabilitation under continuous suprascapular nerve blockade for the treatment of refractory adhesive shoulder capsulitis. Case series. Rev Esp Anestesiol Reanim (Engl Ed). 2022;69(10):625-31.
5. Sa Malheiro N, Afonso NR, Pereira D, Oliveira B, Ferreira C, Cunha AC. [Efficacy of ultrasound guided suprascapular block in patients with chronic shoulder pain: retrospective observational study]. Braz J Anesthesiol. 2020;70(1):15-21.

ELIGIBILITY:
Inclusion Criteria

* Adults aged 18 years or older
* Clinical diagnosis of adhesive capsulitis of the shoulder
* Persistent pain and functional limitation despite initial conservative treatment
* Ability to understand study procedures
* Ability to provide written informed consent

Exclusion Criteria

* Known allergy or hypersensitivity to ropivacaine or methylprednisolone
* Active infection (local or systemic)
* Uncontrolled coagulopathy or ongoing therapeutic anticoagulation
* Recent surgery of the affected shoulder
* Neurological disease affecting the upper limb
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Shoulder Pain - Numeric Rating Scale for Pain (NRS 0-10) | "From enrollment to the end of follow up at 3 years
  Shoulder pain intensity at rest and/or with movement will be measured using the Numerical Rating

CONTACTS AND LOCATIONS:
Locations (1):
- Unidade Local de Saude São João, EPE, Porto, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains sensitive clinical information from a small sample, which may limit the ability to fully de-identify participants while maintaining data integrity. Summary results will be made available through scientific publications and presentations.

REFERENCES:
- [Background] Sa Malheiro N, Afonso NR, Pereira D, Oliveira B, Ferreira C, Cunha AC. [Efficacy of ultrasound guided suprascapular block in patients with chronic shoulder pain: retrospective observational study]. Braz J Anesthesiol. 2020 Jan-Feb;70(1):15-21. doi: 10.1016/j.bjan.2019.11.001. Epub 2020 Feb 19. PMID 32178894
- [Background] Goffin P, Forthomme B, Lecoq JP, Benmouna K, Kaux JF, Fontaine R. Evaluation of intensive rehabilitation under continuous suprascapular nerve blockade for the treatment of refractory adhesive shoulder capsulitis. Case series. Rev Esp Anestesiol Reanim (Engl Ed). 2022 Dec;69(10):625-631. doi: 10.1016/j.redare.2021.06.005. Epub 2022 Nov 4. PMID 36344404
- [Background] Wang JC, Tsai PY, Hsu PC, Huang JR, Wang KA, Chou CL, Chang KV. Ultrasound-Guided Hydrodilatation With Triamcinolone Acetonide for Adhesive Capsulitis: A Randomized Controlled Trial Comparing the Posterior Glenohumeral Recess and the Rotator Cuff Interval Approaches. Front Pharmacol. 2021 May 7;12:686139. doi: 10.3389/fphar.2021.686139. eCollection 2021. PMID 34025441
- [Background] Konarski A, Narayanasamy K, Coghlan J, Chung T, Andrews M, Bell S. A Double Blind Randomised Controlled Trial Comparing Glenohumeral Cortisone With and Without Hydrodilatation in Patients With Frozen Shoulder. ANZ J Surg. 2025 Oct;95(10):2162-2170. doi: 10.1111/ans.70200. Epub 2025 Jun 11. PMID 40495621
- [Background] Brindisino F, Garzonio F, Turolla A, Andriesse A, Pulina F, Cucchi D, Struyf F, Venturin D. Perspectives, perceptions, and expectations of subjects with frozen shoulder: a web-based Italian survey. Arch Physiother. 2024 Dec 9;14:116-130. doi: 10.33393/aop.2024.3244. eCollection 2024 Jan-Dec. PMID 39660343

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-01-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT07380087/Prot_SAP_000.pdf